CLINICAL TRIAL: NCT02128113
Title: A Multicenter, Randomized, Double-Masked, Vehicle-Controlled, Parallel-Group, Phase 2 Study of the Efficacy and Safety of RTA 408 For the Prevention of Corneal Endothelial Cell Loss in Patients Undergoing Cataract Surgery
Brief Title: RTA 408 Ophthalmic Suspension for the Prevention of Corneal Endothelial Cell Loss Following Cataract Surgery - GUARD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RTA 408-C-1309
Record Dates: First submitted 2014-04-28; First posted 2014-05-01 (Estimated); Results first posted 2023-05-26 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Corneal Endothelial Cell Loss; Ocular Pain; Ocular Inflammation; Cataract Surgery
Keywords: RTA 408; Cataract surgery; Corneal Endothelial Cells; omaveloxolone
MeSH Terms: conditions — Corneal Endothelial Cell Loss; Eye Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vehicle Ophthalmic Solution (Placebo Comparator): A single drop of Vehicle Ophthalmic solution was instilled into the study eye twice daily (approximately 12 hours apart) for a maximum of 28 days, beginning 3 to 7 days prior to cataract surgery and continuing on the day of surgery and for 3 weeks after surgery
  Interventions: Drug: Vehicle Ophthalmic Solution
- Omaveloxolone Opthalmic Suspension 0.5% (Experimental): A single drop of Omaveloxolone Ophthalmic suspension 0.5% was instilled into the study eye twice daily (approximately 12 hours apart) for a maximum of 28 days, beginning 3 to 7 days prior to cataract surgery and continuing on the day of surgery and for 3 weeks after surgery
  Interventions: Drug: Omaveloxolone Ophthalmic Suspension 0.5%
- Omaveloxolone Opthalmic Suspension 1% (Experimental): A single drop of Omaveloxolone Ophthalmic suspension 1.0% was instilled into the study eye twice daily (approximately 12 hours apart) for a maximum of 28 days, beginning 3 to 7 days prior to cataract surgery and continuing on the day of surgery and for 3 weeks after surgery
  Interventions: Drug: Omaveloxolone Ophthalmic Suspension 1%

INTERVENTIONS:
Drug: Vehicle Ophthalmic Solution — Opthalmic suspension manufactured to mimic RTA 408 suspension
  Arms: Vehicle Ophthalmic Solution
Drug: Omaveloxolone Ophthalmic Suspension 0.5% — 0.5% ophthalmic suspension of RTA 408
  Other Names: RTA 408 Ophthalmic Suspension 0.5%
  Arms: Omaveloxolone Opthalmic Suspension 0.5%
Drug: Omaveloxolone Ophthalmic Suspension 1% — 1% ophthalmic suspension of RTA 408
  Other Names: RTA 408 Ophthalmic Suspension 1%
  Arms: Omaveloxolone Opthalmic Suspension 1%

SUMMARY:
This study assesses the efficacy and safety of two concentrations of omaveloxolone (RTA 408) ophthalmic suspension for the prevention of corneal endothelial cell loss following cataract surgery.

DETAILED DESCRIPTION:
Many ocular diseases are characterized by oxidative stress and/or inflammation. Oxidative stress is also known to adversely impact corneal endothelial cells, and may be a factor resulting in the acute decrease in corneal endothelial cell density following ocular surgery. While corticosteroids provide potent anti-inflammatory efficacy in a wide range of acute and chronic inflammatory ocular diseases, their use is limited by their side effect profile, which includes the potential to elevate IOP and induce cataract formation. In addition, most available ophthalmic anti-inflammatory treatments, including corticosteroids, do not directly protect against the underlying oxidative stress component of the disease process. Consequently, there is a clinical need for agents that protect against oxidative stress and provide anti-inflammatory efficacy without inducing steroid-like side effects.

This study will assess the safety and efficacy of omaveloxolone (RTA 408) Ophthalmic Suspension (0.5% or 1%) versus vehicle for the prevention of corneal endothelial cell loss in patients undergoing cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Be male or female and ≥18 years of age and ≤80 years of age
2. Plan to undergo cataract extraction by phacoemulsification with the implantation of a posterior chamber intraocular lens
3. Have the potential, in the opinion of the investigator, to improve best-corrected visual acuity in the study eye after surgery
4. Have Grade 3, 4, or 5 nuclear cataract in the study eye, according to the LOCS III
5. Have corneal endothelium in the study eye that can be accurately assessed using specular microscopy
6. Have endothelial cell density of >1800 cells/mm2 in the study eye at the Screening Visit
7. Have a pinhole visual acuity (VA) of at least 1.0 logarithm of the minimum angle of resolution (logMAR) in the study eye and fellow eye as measured using an Early Treatment for Diabetic Retinopathy Study (ETDRS) chart

Exclusion Criteria:

1. Have a score >0 on the ocular pain assessment at the Screening Visit or the Randomization Visit in the study eye
2. Have an active immunosuppressive disease or an autoimmune disease that, in the opinion of the investigator, could affect the quality of the ocular surface
3. Have active or chronic/recurrent ocular or systemic disease that is uncontrolled and will likely affect wound healing
4. Have an intraocular pressure (IOP) ≤5 mmHg in either eye
5. Have had corneal or retinal surgery (laser or incisional) within the past 6 months, or be planning to have laser or incisional surgery during the study period in the study eye
6. Have the presence of guttae Stage 2 or greater or other abnormality in the study eye that does not allow for accurate corneal endothelial cell assessments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2014-05-31 (Actual); Primary Completion 2015-02-28 (Actual); Study Completion 2015-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Harvard Eye Associates, Laguna Hills, California
  - Hull Eye Center, Lancaster, California
  - Argus Research, Cape Coral, Florida
  - Levenson Eye Associates, Jacksonville, Florida
  - Chicago Cornea Consultants, Hoffman Estates, Illinois
  - JacksonEye, Lake Villa, Illinois
  - Discover Vision Centers, Leawood, Kansas
  - Opthalmic Consultants of Boston, Waltham, Massachusetts
  - Talamo Hatch Laser Eye Consultants, Waltham, Massachusetts
  - Associated Eye Care, Stillwater, Minnesota
  - Comprehensive Eye Care, Washington, Missouri
  - Alterman, Modi and Wolter, Poughkeepsie, New York
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - R & R Eye Research, San Antonio, Texas
  - See Clearly Vision Group, McLean, Virginia

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vehicle Ophthalmic Solution | Omaveloxolone Opthalmic Suspension 0.5% | Omaveloxolone Opthalmic Suspension 1%
Started | 103 | 102 | 102
Completed | 100 | 99 | 101
Not Completed | 3 | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Surgery cancelled | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population (all randomized patients)
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle Ophthalmic Solution | Omaveloxolone Opthalmic Suspension 0.5% | Omaveloxolone Opthalmic Suspension 1% | Total
Number analyzed (Participants) | 103 | 102 | 102 | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (7.9) | 67.8 (8.48) | 68.2 (7.44) | 68.4 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 63 | 55 | 170
  Male | 51 | 39 | 47 | 137
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 11 | 9 | 28
  Not Hispanic or Latino | 95 | 91 | 93 | 279
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 3 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 11 | 8 | 24
  White | 95 | 90 | 93 | 278
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 103 | 102 | 102 | 307
Central corneal endothelial cell counts at screening [Mean (Standard Deviation); unit: cell/mm^2] | 2564.4 (329.89) | 2555.7 (342.8) | 2589.6 (332.24) | 2569.9 (334.22)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Central Corneal Endothelial Cell Counts
Description: Count of central corneal endothelial cells 12 weeks post cataract surgery, compared to baseline
Time Frame: 12 weeks
Population: Intent-to-treat population (all randomized patients)
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | Vehicle Ophthalmic Solution | Omaveloxolone Opthalmic Suspension 0.5% | Omaveloxolone Opthalmic Suspension 1%
Number analyzed (Participants) | 98 | 94 | 101
cells/mm^2 | -243.4 (340.58) | -184.8 (237.00) | -260.3 (304.58)
Statistical Analysis 1: Comparison: Vehicle Ophthalmic Solution vs Omaveloxolone Opthalmic Suspension 0.5% vs Omaveloxolone Opthalmic Suspension 1%; Comparison of Omaveloxolone Ophthalmic Suspension pooled (0.5% and 1.0%) versus Vehicle Ophthalmic Solution; Test type: Superiority; p = 0.4529, ANCOVA; Missing data were imputed; LS Mean difference (Net) = 26.95 — Difference is Omaveloxolone Ophthalmic Suspension (pooled) - Vehicle Ophthalmic Solution
Statistical Analysis 2: Comparison: Vehicle Ophthalmic Solution vs Omaveloxolone Opthalmic Suspension 0.5%; Comparison of Omaveloxolone Ophthalmic Suspension 0.5% versus Vehicle Ophthalmic Solution; Test type: Superiority; p = 0.1276, ANCOVA; Missing data were imputed; LS Mean difference (Net) = 64.31 — Difference is Omaveloxolone Ophthalmic Suspension 0.5% - Vehicle Ophthalmic Solution
Statistical Analysis 3: Comparison: Vehicle Ophthalmic Solution vs Omaveloxolone Opthalmic Suspension 1%; Comparison of Omaveloxolone Ophthalmic Suspension 1.0% versus Vehicle Ophthalmic Solution; Test type: Superiority; p = 0.7996, ANCOVA; Missing data were imputed; LS Mean difference (Net) = -11.08 — Difference is Omaveloxolone Ophthalmic Suspension 1.0% - Vehicle Ophthalmic Solution

2. Secondary Outcome: Percentage of Patients With Absence of Anterior Chamber Cells at 2 Weeks After Cataract Surgery
Description: Absence of of anterior chamber cells is defined as anterior chamber cells = 0
Time Frame: 2 weeks
Population: Modified intent-to-treat population (all randomized patients with no imputation for missing data)
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Ophthalmic Solution | Omaveloxolone Opthalmic Suspension 0.5% | Omaveloxolone Opthalmic Suspension 1%
Number analyzed (Participants) | 99 | 98 | 99
Participants
  No | 28 | 41 | 43
  Yes | 71 | 57 | 56
Statistical Analysis 1: Comparison: Vehicle Ophthalmic Solution vs Omaveloxolone Opthalmic Suspension 0.5%; Comparison of Omaveloxolone Ophthalmic Suspension 0.5% versus Vehicle Ophthalmic Solution; Test type: Superiority; p = 0.0647, Cochran-Mantel-Haenszel; Difference in proportion of patients = -13.55, 95% CI 2-sided [-26.75 to -0.36] — Difference is Omaveloxolone Ophthalmic Suspension 0.5% - Vehicle Ophthalmic Solution
Statistical Analysis 2: Comparison: Vehicle Ophthalmic Solution vs Omaveloxolone Opthalmic Suspension 1%; Comparison of Omaveloxolone Ophthalmic Suspension 1.0% versus Vehicle Ophthalmic Solution; Test type: Superiority; p = 0.0517, Cochran-Mantel-Haenszel; Difference in proportion of patients = -15.15, 95% CI 2-sided [-28.34 to -1.96] — Difference is Omaveloxolone Ophthalmic Suspension 1.0% - Vehicle Ophthalmic Solution

3. Secondary Outcome: Percentage of Patients With Absence of Anterior Chamber Flare at 2 Weeks After Cataract Surgery
Description: Absence of of anterior chamber flare is defined as anterior chamber flare = 0
Time Frame: 2 weeks
Population: Modified intent-to-treat population (all randomized patients with no imputation for missing data)
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Ophthalmic Solution | Omaveloxolone Opthalmic Suspension 0.5% | Omaveloxolone Opthalmic Suspension 1%
Number analyzed (Participants) | 99 | 98 | 99
Participants
  No | 11 | 11 | 14
  Yes | 88 | 87 | 85
Statistical Analysis 1: Comparison: Vehicle Ophthalmic Solution vs Omaveloxolone Opthalmic Suspension 0.5%; Comparison of Omaveloxolone Ophthalmic Suspension 0.5% versus Vehicle Ophthalmic Solution; Test type: Superiority; p = 0.9258, Cochran-Mantel-Haenszel; Difference in proportion of patients = -0.11, 95% CI 2-sided [-8.91 to 8.68] — Difference is Omaveloxolone Ophthalmic Suspension 0.5% - Vehicle Ophthalmic Solution
Statistical Analysis 2: Comparison: Vehicle Ophthalmic Solution vs Omaveloxolone Opthalmic Suspension 1%; Comparison of Omaveloxolone Ophthalmic Suspension 1.0% versus Vehicle Ophthalmic Solution; Test type: Superiority; p = 0.6547, Cochran-Mantel-Haenszel; Difference in proportion of patients = -3.03, 95% CI 2-sided [-12.27 to 6.21] — Difference is Omaveloxolone Ophthalmic Suspension 1.0% - Vehicle Ophthalmic Solution

4. Secondary Outcome: Percentage of Patients With Clinical Cure (Absence of Anterior Chamber Cells + Flare) at 2 Weeks After Cataract Surgery
Description: Absence of of anterior chamber cells + flare is defined as anterior chamber cells + flare = 0
Time Frame: 2 weeks
Population: Modified intent-to-treat population (all randomized patients with no imputation for missing data)
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Ophthalmic Solution | Omaveloxolone Opthalmic Suspension 0.5% | Omaveloxolone Opthalmic Suspension 1%
Number analyzed (Participants) | 99 | 98 | 99
Participants
  No | 29 | 42 | 44
  Yes | 70 | 56 | 55
Statistical Analysis 1: Comparison: Vehicle Ophthalmic Solution vs Omaveloxolone Opthalmic Suspension 0.5%; Comparison of Omaveloxolone Ophthalmic Suspension 0.5% versus Vehicle Ophthalmic Solution; Test type: Superiority; p = 0.0657, Cochran-Mantel-Haenszel; Difference in proportion of patients = -13.56, 95% CI 2-sided [-26.84 to -0.28] — Difference is Omaveloxolone Ophthalmic Suspension 0.5% - Vehicle Ophthalmic Solution
Statistical Analysis 2: Comparison: Vehicle Ophthalmic Solution vs Omaveloxolone Opthalmic Suspension 1%; Test type: Superiority — Comparison of Omaveloxolone Ophthalmic Suspension 1.0% versus Vehicle Ophthalmic Solution; p = 0.0526, Cochran-Mantel-Haenszel; Difference in proportion of patients = -15.15, 95% CI 2-sided [-28.42 to -1.88] — Difference is Omaveloxolone Ophthalmic Suspension 1.0% - Vehicle Ophthalmic Solution

5. Secondary Outcome: Percentage of Patients Who Were Pain Free 1 Day After Cataract Surgery
Time Frame: 1 day
Population: Modified intent-to-treat population (all randomized patients with no imputation for missing data)
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Ophthalmic Solution | Omaveloxolone Opthalmic Suspension 0.5% | Omaveloxolone Opthalmic Suspension 1%
Number analyzed (Participants) | 100 | 100 | 102
Participants
  No | 19 | 19 | 18
  Yes | 81 | 81 | 84
Statistical Analysis 1: Comparison: Vehicle Ophthalmic Solution vs Omaveloxolone Opthalmic Suspension 0.5%; Comparison of Omaveloxolone Ophthalmic Suspension 0.5% versus Vehicle Ophthalmic Solution; Test type: Superiority; p = 0.8771, Cochran-Mantel-Haenszel; Difference in proportion of patients = 0.00, 95% CI 2-sided [-10.87 to 10.87] — Difference is Omaveloxolone Ophthalmic Suspension 0.5% - Vehicle Ophthalmic Solution
Statistical Analysis 2: Comparison: Vehicle Ophthalmic Solution vs Omaveloxolone Opthalmic Suspension 1%; Comparison of Omaveloxolone Ophthalmic Suspension 1.0% versus Vehicle Ophthalmic Solution; Test type: Superiority; p = 0.8248, Cochran-Mantel-Haenszel; Difference in proportion of patients = 1.35, 95% CI 2-sided [-9.32 to 12.02] — Difference is Omaveloxolone Ophthalmic Suspension 1.0% - Vehicle Ophthalmic Solution

6. Secondary Outcome: Change From Baseline in Central Corneal Endothelial Cell Counts
Description: Count of central corneal endothelial cells 6 weeks post cataract surgery, compared to baseline
Time Frame: 6 weeks
Population: Intent-to-treat population (all randomized patients)
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | Vehicle Ophthalmic Solution | Omaveloxolone Opthalmic Suspension 0.5% | Omaveloxolone Opthalmic Suspension 1%
Number analyzed (Participants) | 94 | 96 | 98
cells/mm^2 | -238.2 (344.73) | -193.9 (269.54) | -242.2 (291.14)
Statistical Analysis 1: Comparison: Vehicle Ophthalmic Solution vs Omaveloxolone Opthalmic Suspension 0.5% vs Omaveloxolone Opthalmic Suspension 1%; Comparison of Omaveloxolone Ophthalmic Suspension pooled (0.5% and 1.0%) versus Vehicle Ophthalmic Solution; Test type: Superiority; p = 0.4686, ANCOVA; Missing data were imputed; LS Mean difference (Net) = 27.21
Statistical Analysis 2: Comparison: Vehicle Ophthalmic Solution vs Omaveloxolone Opthalmic Suspension 0.5%; Comparison of Omaveloxolone Ophthalmic Suspension 0.5% versus Vehicle Ophthalmic Solution; Test type: Superiority; p = 0.2636, ANCOVA; Missing data were imputed; LS Mean difference (Net) = 49.99
Statistical Analysis 3: Comparison: Vehicle Ophthalmic Solution vs Omaveloxolone Opthalmic Suspension 1%; Comparison of Omaveloxolone Ophthalmic Suspension 1.0% versus Vehicle Ophthalmic Solution; Test type: Superiority; p = 0.9691, ANCOVA; Missing data were imputed; LS Mean difference (Net) = -1.74

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Investigators reported all AEs and SAEs that were observed or reported by patients from the time of first dose until the final visit, regardless of their relationship to study drug or their clinical significance.
Arm/Group | Vehicle Ophthalmic Solution | Omaveloxolone Opthalmic Suspension 0.5% | Omaveloxolone Opthalmic Suspension 1%
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/102 | 0/102
Serious Adverse Events (participants affected / at risk) | 4/103 | 0/102 | 4/102
Other Adverse Events (participants affected / at risk) | 27/103 | 33/102 | 36/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Ophthalmic Solution (N=103) | Omaveloxolone Opthalmic Suspension 0.5% (N=102) | Omaveloxolone Opthalmic Suspension 1% (N=102)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Ophthalmic Solution (N=103) | Omaveloxolone Opthalmic Suspension 0.5% (N=102) | Omaveloxolone Opthalmic Suspension 1% (N=102)
Anterior chamber inflammation (Eye disorders) | 2 (2) | 3 (3) | 3 (3)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 4 (4) | 5 (5)
Eye inflammation (Eye disorders) | 2 (2) | 4 (4) | 3 (3)
Eye irritation (Eye disorders) | 0 (0) | 4 (4) | 6 (6)
Eye pain (Eye disorders) | 4 (5) | 6 (6) | 4 (4)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 4 (4) | 4 (4)
Lacrimation increased (Eye disorders) | 1 (1) | 5 (5) | 9 (10)
Ocular hyperaemia (Eye disorders) | 0 (0) | 3 (3) | 4 (4)
Ocular hypertension (Eye disorders) | 5 (6) | 8 (9) | 5 (5)
Photophobia (Eye disorders) | 3 (3) | 3 (3) | 8 (8)
Posterior capsule opacification (Eye disorders) | 5 (5) | 9 (10) | 3 (4)
Punctate keratitis (Eye disorders) | 3 (4) | 4 (4) | 4 (5)
Cataract operation complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Intraocular pressure increased (Investigations) | 7 (7) | 1 (1) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.